CLINICAL TRIAL: NCT04224220
Title: Effectiveness of Nurse-based Care Coordination on Readmissions Among Primary Care Patients: a Stepped Wedge Cluster Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michelle A. Lampman, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-009784
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Patient Activation
MeSH Terms: conditions — Patient Participation | interventions — Remote Patient Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Adult Medical Care Coordination (Active Comparator): This group will receive adult medical care coordination following discharge from a recent hospitalization.
  Interventions: Other: Adult Medical Care Coordination
- Remote Patient Monitoring (Active Comparator): This group will receive remote patient monitoring following discharge from a recent hospitalization.
  Interventions: Other: Remote Patient Monitoring
- Usual Care (No Intervention): The usual care group will not receive additional supportive care following discharge from a recent hospitalization beyond what is typically offered through their primary care team.

INTERVENTIONS:
Other: Adult Medical Care Coordination — Nurse-based support that includes a home visit and follow-up coaching telephone calls to monitor patient status and ability to self-manage symptoms.
  Arms: Adult Medical Care Coordination
Other: Remote Patient Monitoring — Nurse-based support and coaching that incorporates the use of technology to monitor patient status and ability to self-manage symptoms.
  Arms: Remote Patient Monitoring

SUMMARY:
This trial will evaluate the effectiveness of nurse-based care coordination and nurse-based remote patient monitoring on hospital readmissions among primary care patients.

ELIGIBILITY:
Inclusion Criteria:

* Discharged from the hospital in the past 7 days
* LACE+ score of 59 or greater and at least two chronic conditions
* Index hospitalization with discharge directly to community dwelling home (home, assisted living)
* English speaking
* Normal cognitive function - mild dementia or mild cognitive impairment is allowed if a caregiver is able to work with the care coordinator and patient during program enrollment
* Mayo Clinic or Mayo Clinic Health System provider managing the patient's care (e.g. primary care); patient is assigned to the panel of a Mayo Clinic Medical Doctor/Nurse Practitioner/Physician Assistant
* Access to and ability to communicate via telephone (either patient or caregiver)

Exclusion Criteria:

* Psychiatric hospital admission
* Patients with a serious and persistent mental health disorder or severe treatment interfering behavior that require a higher level of service than is available at the patient's clinic
* Untreated active substance or alcohol abuse
* Dementia or moderate to severe cognitive impairment
* Discharged to one of the following: rehabilitation unit, skilled nursing facility, assisted living memory unit, group home
* Pregnancy
* Active treatment for cancer
* Receiving dialysis or transplant services
* Life expectancy < 6 months or enrolled in hospice or palliative care programs
* Patient is unwilling to sign a Release of Information (ROI); ROI allows those providing care, internal and external, to be actively involved in the patient's care coordination
* Patients with active tuberculosis (TB)
* Violent patient flag noted in Epic (for adult medical care coordination)
* Patient declines home visit (for adult medical care coordination)
* Patient is already enrolled in remote patient monitoring or the care transitions program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1947 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Rate of Readmission | 30 days
  The rate of patients revisiting the emergency department or being admitted to the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Lampman, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials